CLINICAL TRIAL: NCT00160472
Title: Evaluation of Vasopressin and Vasopressin Receptor Expression in the Arteries and Veins of Ovarian Neoplasms
Brief Title: Evaluation of Vasopressin in the Vessels of Ovarian Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Organization: Tripler Army Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TAMC 3H04
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2004-03

CONDITIONS: Ovarian Neoplasms
Keywords: vasopressin; ovarian; neoplasm
MeSH Terms: conditions — Ovarian Neoplasms; Diabetes Insipidus; Neoplasms

INTERVENTIONS:
Procedure: removal of ovarian vessels

SUMMARY:
This study will evaluate the expression of arginine vasopressin (AVP) by peptide and mRNA quantitation and also measurement of its V1 receptor mRNA, in the arteries and veins of ovarian malignant (cancerous) or benign (non-cancerous) tissue. The investigators will examine whether AVP protein and AVP and V1 receptor mRNA expression vary with respect to tumor histology, intratumoral vascularization and systemic blood pressure.

DETAILED DESCRIPTION:
d. STATUS: Background and Significance/Preliminary Studies

Neovascularization is an obligate early event in cancer growth. Consequently, angiogenesis appears to play an important role in disease progression and survival of most malignancies in general and gynecologic malignancies specifically. Ovarian cancer is the second most common gynecologic malignancy, and the leading cause of cancer related death among the gynecologic malignancies. It is estimated that 23,300 new cases of ovarian cancer will be diagnosed in the United States in 2003 and that 13,900 women will die from disease. Angiogenesis may serve as a prognostic indicator in ovarian cancer. Angiogenesis in cancer requires the proliferation and migration of endothelial cells in response to a variety of cytokines to include angiogenin, endothelial cell growth factor, and vascular endothelial growth factor (VEGF). The expression of some of these cytokines have been evaluated in gynecologic malignancies. Increased expression of VEGF protein by immunohistochemistry has been associated with decreased disease free survival 18 versus 120 months in early stage epithelial ovarian cancers. Conversely any exposure to antiangiogenic factors should inhibit tumor cell growth in vitro. Angiostatin and endostatin have also been found to inhibit ovarian cancer growth in mice 7.

The neovascularization required of fast growing malignancies in general, and ovarian cancer specifically, necessitates that they contain many new vessels that have less smooth muscle in their walls. Because of the quantitative decrease in vascular smooth muscle these vessels also have a decreased resistance to blood flow than the vessels found in benign tumors. Malignant tumors with low vascular resistance have been shown to demonstrate decreased smooth muscle actin expression and intense Cd34 expression with no differences in microvessel density (MVD) noted 8. Immunohistochemical analysis using monoclonal antibodies against smooth muscle actin (SMA) and CD34 (an endothelial cell marker) demonstrated that low resistance to blood flow in vessels within malignant ovarian tumors may be associated with a poorly developed muscular coat in the tumor vessels, compared with that observed in benign tumors. Color-flow Doppler imaging uses the altered blood flow patterns as a marker in an attempt to differentiate benign from malignant tumors 9. Researchers have evaluated the presence of intratumoral vascularization in ovarian neoplasms by Color-flow Doppler ultrasound. Benign tumors and cysts have a significantly higher pulsatility index (PI) (mean, 1.93 +/- 1.02; range, 0.23-3.99) and resistive index (RI) (mean, 0.77 +/- 0.22; range, 0.2-1.0) than do malignant tumors (PI: mean, 0.77 +/- 0.33; range, 0.31-1.09; RI: mean, 0.5 +/- 0.17; range, 0.27-0.67). Some overlap, however, exists in individual values for benign and malignant lesions. The difference in the angiogenic and vascular resistant natures of benign and malignant ovarian tumors showing intratumoral blood flow may thus be correlated with the endothelial cell activity of the tumor vessels and not the MVD. This low resistance to blood flow within tumor vessels and subsequent endothelial cell activity could be regulated by local, endothelial cell or vascular smooth muscle cell, arginine-vasopressin (AVP) synthesis and release with subsequent actions on vasopressin receptors.

Arginine-vasopressin (AVP) is a peptide hormone classically known to be synthesized in the hypothalamus and secreted by the posterior pituitary gland. AVP has a variety of roles in the body and a variety of systemic physiologic functions to include vasoconstriction, gluconeogenesis, corticosteroidogenesis, and excretion of water and urea. AVP causes a peripheral vasoconstriction that is thought to be mediated primarily by the V1 receptor. AVP is thought to do this by a variety of mechanisms to include activation of the V1a receptors with stimulation of phospholipase A2 which leads to increased calcium spiking activity. AVP could also do this by regulating the expression of other hypertensive factors and proteins in the body. AVP has been shown to play an important role in the development of hypertension following aortic constriction in rats. When rats were given AVP following constriction of the abdominal aorta, hypertension developed and these animals had an increased response to angiotensin II. Therefore AVP is thought to permit the expression of other factors such as angiotensin II. The presence of AVP is important in other animal models of hypertension such the spontaneously hypertensive rat and DOCA salt hypertension. For instance, administration of DOCA salt to Brattleboro rats, genetically incapable of synthesizing vasopressin in the hypothalamus, will not result in the development of hypertension. However, with administration of exogenous AVP, these rats will develop hypertension when given DOCA salt treatment.

Exposure of vascular smooth muscle cells to AVP also increases smooth muscle actin through activation of all three MAP kinase family pathways. Because AVP has the ability to regulate and increase smooth muscle actin this suggests that AVP may not only regulate growth of vascular smooth muscle but also promote expression of smooth muscle-specific contractile proteins . Previous studies have shown that AVP can produce an exaggerated vascular vasoconstriction in young spontaneously hypertensive rats (SHR) relative to normotensive rats. This exaggerated response was likely associated to a higher density of V1 receptors associated with increased AVP gene expression. Finally AVP and other neuropepetides have been shown to serve as autocrine growth factors for some solid tumors. The mitogenic influence of AVP is thought to involve increases in intracellular calcium. AVP is often expressed in small cell lung cancer (SCLC), and can act as an autocrine growth factor in these cancers. AVP expression in SCLC is thought to be dependent on the modulation of normal repressor activity 12. Because AVP has been implicated in the physiology of vascular constriction and mean vascular pressure, and also because it has been shown to be expressed in certain types of cancer, it may also have a role as an angiogenic factor in intratumoral vascularization in ovarian cancer carcinogenesis. It is the purpose of our proposed study to investigate the relationship between AVP expression and its vascular receptor with ovarian neoplasm histology.

Preliminary results:

Recently, our labs have isolated and analyzed human mesenteric arteries for VP mRNA and V1 receptor mRNA analyses. V1R mRNA was strongly positively correlated with diastolic blood pressure (r = 0.70, p = 0.0112). V1R mRNA tended to be greater in males than females (5.73 + 1.29 compared to 2.3 + 0.94 relative expression units of V1R mRNA, p = 0.057). Also, arterial AVP mRNA correlated negatively with age (p=0.0028). These results suggest that alterations in both VP and V1R expression could be involved in disease states such as ovarian cancer where blood pressure and flow as well as age may be factors in the development of the malignancy of the tumor.

The AVP peptide was measured by radioimmunoassay in other blood vessels23, e.g. radial and mammary artery and saphenous vein samples, and the immunoactivity was shown to co-migrate with synthetic AVP on HPLC analysis. The levels of hormone ranged from undetectable to as high as 60 uU/gr tissue. Thus, we will also be able to verify changes in VP gene expression by measuring the AVP protein directly in the ovarian neoplasm blood vessels collected.

6. PLAN: Women, 18 years old or greater, who are having their ovaries removed will be enrolled in the protocol. 110 total specimens will be obtained. At our institution approximately 200 patients per year have ovaries removed. All patients who have had gynecologic tissue removed for benign (non cancerous) or malignant (cancerous) indications will meet inclusion criteria. Patients who have a malignancy that is not a primary gynecologic malignancy will be excluded from the study. Each patient's intratumoral vascularity will be assessed by Doppler ultrasound and systemic blood pressure measured preoperatively.

PROCEDURE FOR PROCUREMENT, PREPARATION AND SHIPMENT OF TISSUE SPECIMENS Ovarian arterial and venous specimens will be collected for analysis of AVP peptide and for AVP and vasopressin receptor mRNA. Operating room personnel will be asked to keep the tissue, ovarian artery and vein segments, fresh and not put it in fixative. Promptly following removal of the tissue, the specimens will be prepared as follows: The most sterile primary tissue will be cut to measure at least 5.0 cm in length. The tumor tissue will then be separated from as much connective tissue as possible. The specimen will be placed in the RNA preservative RNAlaterTM, placed on wet ice and sent to the Department of Clinical Investigation Laboratories quickly. Laboratory analyses of AVP peptide and for AVP and vasopressin receptor mRNA isolation and quantitation will be performed in the Physiology and Research Pharmacology laboratories of the Department of Clinical Investigation.

Laboratory Methods: Vasopressin synthesis (as indicated by VP mRNA) and vasopressin receptor (V1R or V2R) up or down regulation (as indicated by V1R mRNA or V2R mRNA levels) will be assessed. Measurement of V2R in addition to V1R mRNA will help clarify whether possible changes in V1R expression in the ovarian neoplasms are specific to that receptor subtype. Ovarian artery samples will be isolated and stored in RNA later TM (Ambion, Austin, TX) at -70oC until extracted for RNA with a commercial kit (Invitrogen Carlsbad, CA). VP mRNA, V1R mRNA, and beta actin mRNA will be quantified by quantitative real-time PCR (qPCR) using an iCycler (BioRad Laboratories, Hercules, CA). Reverse transcription of the RNA to cDNA will be done using Superscript TM (Invitrogen), and PCR will be done with Platinum qPCR SuperMix-UDG (Invitrogen). Standard curves will be generated using dilutions of a stock of human blood vessel cDNA and the cycle threshold for each sample will be related to a dilution's assigned copy number. qPCR data will be expressed as a ratio of VP, V1R, or V2R mRNA copies per beta-actin mRNA copies. Product generation on all three mRNA segments we are measuring, yield slopes of approximately 3.3 indicating nearly 100% efficiency of a doubling of product with each cycle in temperature, and gel electrophoresis indicates one band of product. All quantitation is done through the detection of increasing intensity of a specific fluorescent probe for each product.

Vasopressin peptide will be analyzed by radioimmunoassay of vascular tissue extracts. The tissue will be extracted by first rinsing the tissue free of blood with 0.1 N Acetic Acid, blotting and weighing the tissue. The specimen will placed in cold 1.0 N HCl (1ml/0.5 g tissue) and homogenized with a Polytron for 1 min. The homogenate will then be centrifuged at 27,000 G for 45 min. The supernatant will be saved, and the pellet resuspended and rehomogenized in 1 ml 1.0 N HCl, and centrifuged. The supernatants are then combined. The supernatants will then be extracted as routinely done with plasma samples by absorption on to octadecylsilane cartridges (SepPak, C-18, Waters, Milford, MA) and eluted with acidified ethanol. The eluate is dried by vacuum and suspended in assay buffer. At this point the sample can be applied to C-18 HPLC column and eluted in a single phase buffer system consisting of 0.05 M NH4AC in 39% MeOH, and each 1-ml fraction, dried under vacuum, and suspended in radioimmunoassay buffer and assayed. Alternatively, the HPLC fractionation may not have to be done after initial confirmation that no interference is present in the initial sample. In this case, the initial extract will be assayed by radioimmunoassay directly.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had gynecologic tissue removed for benign (noncancerous) or malignant (cancerous) indications.

Exclusion Criteria:

* Patients who have a malignancy that is not a primary gynecologic malignancy.
* Age less than 18
* Males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2004-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Compare the levels of AVP and the vasopressin V1 receptor expression in the arteries and veins of ovarian tissue found to be cancerous versus ovarian tissue found to be noncancerous
Correlate the expression of AVP and its V1 receptor to stage of ovarian neoplasms graded by histology assessment
Correlate the expression of AVP and its receptor to intratumoral vascularization through Doppler ultrasound and systemic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: John H Farley, MD, Principal Investigator — Uniformed Services Unievrsity of the Health Sciences
Locations (1):
- Tripler Army Medical Center, Honolulu, Hawaii, United States